CLINICAL TRIAL: NCT01008020
Title: A Randomized Controlled Study on the Effects of Tea Catechin Consumption on the Prevention of Influenza Infection in Healthy Adults
Brief Title: Effects of Tea Catechin Consumption on the Prophylaxis of Influenza Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masahiro Morikawa (Other)
Collaborators: White Cross Nursing Home (Other)
Responsible Party: Sponsor-Investigator, Masahiro Morikawa, Clinical Trials management office, University of Shizuoka
Organization: University of Shizuoka (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT2009002
Record Dates: First submitted 2009-10-29; First posted 2009-11-05 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Influenza Infection
Keywords: tea catechin extracts; influenza infection; prophylaxis; supplements; adults over 20 years old; both men and women

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement: placebo (No Intervention)
- Tea catechin extracts (Active Comparator)
  Interventions: Dietary Supplement: tea catechin extracts

INTERVENTIONS:
Dietary Supplement: tea catechin extracts — Tea catechin extracts 540 mg/day, are consumed for 5 months.
  Arms: Tea catechin extracts

SUMMARY:
The Purpose of this study is to evaluate the effects of 5 months catechin consumption on the prevention of influenza infection.

DETAILED DESCRIPTION:
Catechins are the major components of tea flavonoids and are reported to possess physiological activities such as antiviral effects. Recent experimental studies have revealed that tea catechin extracts prevent influenza infection, but few studies have been conducted on the clinical effects of tea catechin consumption on the prophylaxis of influenza infection. Based on these backgrounds, we designed a prospective randomized controlled study to evaluate the effects of 5 months tea catechin consumption on the prophylaxis of influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* aged over 20 years
* possible to maintain without drinking tea more than 250 ml per day during the study
* possible to maintain without taking supplements or herbal products including catechin extracts during the study
* possible to fill out a questionnaire personally
* Obtained written informed consent before participation

Exclusion Criteria:

* Possessing some chronic infectious diseases in need of therapy
* Possessing tea or catechin allergy
* Possessing a history of influenza infection before six months prior to the study
* diagnosed as inadequate for other reasons to participate the study by principal investigator

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
the incidence rates of influenza infection | Until 5 months consumption of the study capsules

SECONDARY OUTCOMES:
the incidence rates of upper respiratory tract infections | Until 5 months consumption of the study capsules
the severity of the symptoms and the duration of the cold among incident cases | Until 5 months consumption of the study capsules
occurrence of the adverse events | Until 5 months consumption of the study capsules

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamada, MD, PhD, Study Chair — University of Shizuoka
Locations (1):
- White Cross Nursing Home, Higashimurayama, Tokyo, Japan

REFERENCES:
- [Derived] Matsumoto K, Yamada H, Takuma N, Niino H, Sagesaka YM. Effects of green tea catechins and theanine on preventing influenza infection among healthcare workers: a randomized controlled trial. BMC Complement Altern Med. 2011 Feb 21;11:15. doi: 10.1186/1472-6882-11-15. PMID 21338496